CLINICAL TRIAL: NCT03852706
Title: A Randomized Controlled Pilot Trial of Low-resolution Brain Electromagnetic Tomography (LORETA) Neurofeedback Training for Treatment-resistant Auditory Verbal Hallucinations in Schizophrenia
Brief Title: EEG-based Neurofeedback for Auditory Verbal Hallucinations (HALFEED)
Acronym: HALFEED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A national Covid-19 lockdown prevented completion of the trial
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Actualise (Other)
Responsible Party: Principal Investigator, Simon McCarthy-Jones, Associate Professor in Clinical Psychology and Neuropsychology, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 206789; 25911 (Other Grant/Funding Number: Brain & Behavior Research Foundation)
Record Dates: First submitted 2019-01-25; First posted 2019-02-25 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Schizophrenia
Keywords: Hallucinations
MeSH Terms: conditions — Schizophrenia; Hallucinations | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LORETA (Experimental): In the first session, Low Resolution Brain Electromagnetic Tomography (LORETA) will be used in combination with Z-scores to identify participants' resting state EEG differences relative to a database of norms of their demographic. EEG abnormalities which are consistent with the research literature on neural changes associated with AVH will then be targeted for normalization using neurofeedback training using LORETA in combination with Z-scores.
  Interventions: Other: LORETA; Other: Treatment as usual
- Treatment as usual (Other): Maintenance use of an atypical antipsychotic (e.g., clozapine) with support, when needed, of a community nurse.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: LORETA — Twenty sessions of neurofeedback training using LORETA in combination with z-scores.
  Arms: LORETA
Other: Treatment as usual — Treatment-as-usual

SUMMARY:
This study's primary objective is to perform a randomized controlled pilot study to assess the feasibility of using EEG-based neurofeedback to reduce the severity of treatment-resistant auditory verbal hallucinations ('hearing voices') in patients diagnosed with schizophrenia. Patients will be randomized to receive either EEG-based neurofeedback or treatment-as-usual.

DETAILED DESCRIPTION:
Auditory verbal hallucinations (AVH) are experienced by up to 80% of patients diagnosed with schizophrenia, where they can cause significant occupational and social impairment. Current treatments are incompletely effective. Around 25-30% of AVH are refractory to antipsychotic drugs, and cognitive behavioural therapy only shows a small-medium effect size. Initially promising studies of neurostimulation have shown smaller effect sizes as better controlled trials have been conducted. There is hence the need for innovative new treatments. One potential option is neurofeedback training. The primary objective of study is to perform a randomized, controlled, rater-blinded pilot trial (n=40) of EEG neurofeedback for AVH in patients with treatment-resistant schizophrenia, to assess trial process, which will then inform a future definitive trial. The secondary objective is to calculate a 95% confidence interval that will allow interpretation of statistical difference between neurofeedback and treatment-as-usual groups to assess neurofeedback for reducing auditory verbal hallucinations. Participants will be randomly allocated to either a neurofeedback (plus treatment-as-usual) or treatment-as-usual alone condition. Neurofeedback will employ Z-score based LORETA (Low Resolution Brain Electromagnetic Tomography). After a baseline assessment, twenty sessions of personalized neurofeedback training will be delivered over a period of approximately four months. This is the first registered trial of EEG neurofeedback for hallucinations. The primary focus of the pilot trial is on feasibility. However, a 95% confidence interval will be determined for the difference on PSYRATS-AH and AHRS scores between neurofeedback and treatment-as-usual to help inform a future definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥ 18 years old
* Have a clinical diagnosis of a schizophrenia-spectrum disorder
* Have been experiencing auditory verbal hallucinations for at least one year
* Score 2 or more on the frequency item of the auditory hallucinations subscale of the Psychotic Symptom Ratings Scale (PSYRATS-AH; Haddock et al., 1999) at time of initial assessment (representing voices occurring at least once a day)
* Are deemed refractory to antipsychotic treatment (defined as still hearing voices despite 4-6 weeks of treatment with two different antipsychotics)
* Have been on a stable dose of antipsychotic medication for the three months prior to study enrolment
* Are right-handed, as determined by the Edinburgh Handedness Inventory (Oldfield, 1971)
* Are able to provide written, informed consent.

Exclusion Criteria:

* Having a diagnosed substance abuse disorder
* Prior head injury with loss of consciousness for more than five minutes
* At immediate risk of harm to self or others.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 24 months
  We will measure how many patients were recruited into the trial per calendar month of active recruitment.
Willingness of participants to be randomised. | 24 months
  We will measure the proportion of patients who were entered in the trial but refused randomisation.
Willingness of participants to complete assessments | 24 months
  We will measure the proportion of participants who were entered into the trial and completed all baseline assessment measures.
Drop-out rate: LORETA condition | 24 months
  We will measure the proportion of patients who were entered into the trial, randomised to the neurofeedback condition, and dropped out of the study.
Success of blinding of raters | 24 months
  We will measure the proportion of blind raters who were correctly able to guess the group allocation of participants, and assess if this was greater than chance.
Rates of adverse psychiatric events | 24 months
  We will assess the proportion of patients entered into the trial who experienced adverse psychiatric events reported.
Drop-out rate: Controls | 24 months
  We will measure the proportion of patients who were entered into the trial, randomised to the control condition, and dropped out of the study.

SECONDARY OUTCOMES:
Auditory Hallucination Subscale of the Psychotic Symptom Ratings Scale (PSYRATS-AH) | End of intervention (~4 months)
  The Auditory Hallucination Subscale of the Psychotic Symptom Ratings Scale (PSYRATS-AH; Haddock et al., 1999) is an 11-item measure of the severity of auditory verbal hallucinations. Total scores can range from 0 to 44 with higher scores indicating greater severity of auditory verbal hallucinations. The PSYRATS-AH has been found to have a four-factor structure (Woodward et al., 2014). These are Emotion (range 0-20), Physical (range 0-12), Cognitive (range 0-8) and Loudness (range 0-4). Higher scores on each of these subscales represents more severe auditory verbal hallucinations. We will assess between group differences in both the total and four factor scores of the PSYRATS-AH at end of therapy.
Auditory Hallucinations Rating Scale (AHRS) | End of intervention (~4 months)
  The Auditory Hallucinations Rating Scale (AHRS; Hoffman et al., 2003) is a seven-item structured clinical interview, which assesses the severity of auditory verbal hallucinations in the past week. Its items assess frequency, reality, loudness, number, length, attentional salience (how demanding of attention the voice is) and distress level. Items are rated on unique scales. Total scores on this measure can range from 0 - 41 . Higher scores represent more severe auditory verbal hallucinations.
Delusions Subscale of the Psychotic Symptom Ratings (PSYRATS-D). | End of intervention (~4 months)
  Delusions will be assessed by the Delusions Subscale of the Psychotic Symptom Ratings Scale (PSYRATS-D; Haddock et al., 1999). This is a 6-item structured clinical interview. Total scores can range from 0-24, with higher scores representing more severe delusions. It has been found to have two factors (Woodward et al., 2014), namely Distress (distress amount, distress intensity) and Frequency (preoccupation amount, preoccupation duration, conviction, disruption). Total scores on these factors can range from 0-8 and 0-16 respectively, with higher scores representing more severe delusions. Both total PSYRATS-D and factor scores will be employed.
Hospital Anxiety and Depression scale | End of intervention (~4 months)
  The Hospital Anxiety and Depression scale (HADS; Zigmund & Snaith, 1983) is a 16-item self-report measure of both anxiety and depression. Eight items assess depression and eight items assess anxiety. Depression scores can range from 0-24 with higher scores representing higher levels of depression. Anxiety scores can range from 0-24 with higher scores representing higher levels of anxiety.
Quality of Life Enjoyment and Satisfaction Questionnaire | End of intervention (~4 months)
  Quality of life will be assessed by the short-form of the self-report Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ; Endicott et al., 1993). Total scores on 16-item measure can range from 14 to 70, with higher scores representing greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Simon McCarthy-Jones, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Tallaght University Hospital / St. James' Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No